CLINICAL TRIAL: NCT01876589
Title: Impact of Vascular Reparative Therapy on Vasomotor Function and Myocardial Perfusion: a Randomized H215O PET/CT Study
Brief Title: Impact of Vascular Reparative Therapy on Vasomotor Function and Myocardial Perfusion:a Randomized H215O PET/CT Study
Acronym: VANISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Wynand Stuijfzand, Drs, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VANISH
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease (CAD); Invasive coronary angiography (ICA); Positron Emission Tomography (PET)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable vascular scaffold (Active Comparator): Paritcipants will receive a bioresorbable vascular scaffols (BVS)
  Interventions: Device: Bioresorbable vascular scaffold
- Xience Prime (Active Comparator): Participant will receive a Xience Prime stent
  Interventions: Device: Xience Prime

INTERVENTIONS:
Device: Bioresorbable vascular scaffold — Drug eluting coronary stent, resorbable in 2-3 years
  Arms: Bioresorbable vascular scaffold
Device: Xience Prime — Drug eluting metallic stent
  Arms: Xience Prime

SUMMARY:
The purpose of this study is to examine the improvement of myocardial blood flow induced by regained vasomotor functions of the stented coronary segment after resorption of BVS over time.

DETAILED DESCRIPTION:
Objective The objective of the proposed study is to determine the impact of VRT, in comparison with conventional drug-eluting stenting, on endothelium dependent vasodilation and maximal hyperemic myocardial perfusion using H215O PET.

Study design The study is designed as a single center single-blind randomized clinical trial and will be conducted at the VU University Medical Center in Amsterdam.

Summary of the study design It is hypothesized that VRT will result in augmented endothelium dependent coronary vasodilation and maximal myocardial perfusion as compared with conventional stenting of a coronary lesion. Within one year sixty patients (age 18-65) with documented single vessel CAD (type A or B1 lesion) accepted for PCI based on clinical grounds and according to current international guidelines, will be asked to participate in this trial. Patients will be randomized to implantation of a drug-eluted stent (Xience Prime) or BRS (Absorb). The patients will be blinded to the nature of the implanted device. H2 15O PET will be performed one month (reference scan), one year, and three years after the PCI procedure (resolution of BRS is generally complete within a three year period). The PET protocol will consist of three MBF measurements: resting MBF, during endothelial dependent vasodilation provoked by coldpressor-testing (CPT), and during (endothelial dependent and independent) maximal vasodilation by infusion of adenosine intravenously. After three years a control invasive coronary angiogram will document any potential obstructive coronary lesions that may affect the MBF measurements.

Primary study parameters/outcome of the study MBF measurements: resting MBF, during endothelial dependent vasodilation provoked by cold-pressor-testing (CPT), and during (endothelial dependent and independent) maximal vasodilation by infusion of adenosine intravenously

Secondary study parameters/outcome of the study Obstructive coronary lesions on control invasive coronary angiogram that may affect the MBF measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented obstructive CAD by invasive coronary angiography resulting in myocardial ischemia (either documented by invasive (i.e. fractional flow reserve, FFR) or noninvasive imaging techniques (e.g. exercise ECG, myocardial perfusion imaging, or inducibility of wall motion abnormalities during dobutamine stress).
* Presence of a single, de-novo lesion in a native coronary artery (type A or B1), with a reference vessel diameter of at least 3.0 mm and a diameter stenosis of 50% or more and less than 100%, with a thrombolysis in myocardial infarction (TIMI) flow grade of at least 2. Coronary lesion must be amendable for successful treatment with one of the following BRS device dimensions: length 18 or 28 mm, diameter 3.0 or 3.5 mm.

Exclusion Criteria:

* age of 65 or above
* refusal or inability to provide written informed consent
* other than single CAD
* abnormal echocardiographic findings (i.e. wall motion abnormalities, ventricular hypertrophy, valvular disease etc.)
* complex coronary lesion characteristics (e.g. lesions located in the left main coronary artery, lesions involving a side branch more than 2 mm in diameter, and the presence of thrombus or another clinically significant stenosis in the target vessel)
* poor kidney function defined as an eGFR < 30 ml/min
* astma or chronic obstructive pulmonary disease
* other than sinus rhythm
* pregnancy
* bail out stenting after placement of the study device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Myocardial Blood Flow over time | Three years
  Endothelial dependent vasomotor function and effect on myocardial perfusion

SECONDARY OUTCOMES:
Restenosis | Three years
  Obstructive coronary lesions and lumen dimensions on control invasive coronary angiogram that may affect the MBF measurements

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands